CLINICAL TRIAL: NCT03813069
Title: A Within-subject Laboratory and Field Trial to Test the Use of Commercially Available Insect Repellents Against Contact From Musca Sorbens, the Putative Vector of Trachoma
Brief Title: Testing Insect Repellents Against Musca Sorbens, the Vector of Trachoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Federal Minstry of Health of Ethiopia (Other Government); Oromia Regional Health Bureau, Ethiopia (Unknown); The Fred Hollows Foundation, Ethiopia (Unknown); The Fred Hollows Foundation, UK (Unknown); The Fred Hollows Foundation, Australia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-kep-132
Record Dates: First submitted 2019-01-07; First posted 2019-01-23 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Trachoma
MeSH Terms: conditions — Trachoma | interventions — ethyl-3-(N-n-butyl-N-acetyl)aminopropionate; Permethrin

STUDY DESIGN:
Intervention Model Description: This is a within-subject, non-masked, trial of the use of commercially available insect repellents against Musca sorbens, with two consecutive participant groups in the laboratory and in the field, and a primary endpoint of measuring the protective efficacy of each repellent product.
  The first (laboratory-based) study has one arm, in which all participants test all repellent products. Those that are found to generate at least 30 % protective efficacy will be tested in the second (field-based) study, which will have four arms. Up to three arms will test a repellent product and there will be a control arm.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Laboratory study (Other)
  Interventions: Other: IR3535; Other: Permethrin lower dose; Other: Permethrin higher dose
- Field study: IR3535 (Other)
  Interventions: Other: IR3535
- Field study: Permethrin lower dose (Other)
  Interventions: Other: Permethrin lower dose
- Field study: Permethrin higher dose (Other)
  Interventions: Other: Permethrin higher dose
- Field study: control arm (No Intervention)

INTERVENTIONS:
Other: IR3535 — The topical repellent IR3535 (3-[N-butyl-N-acetyl]-aminopropionic acid ethyl ester) only
  Arms: Field study: IR3535; Laboratory study
Other: Permethrin lower dose — A fabric scarf, impregnated with the insecticide permethrin (m-Phenoxybenzyl)-cis,trans-3-(2,2-dichlorovinyl)-2,2-dimethylcyclopropanecarboxylate) that has contact irritancy/spatial repellency. Dose appropriate to children of 10-20 kg.
  Arms: Field study: Permethrin lower dose; Laboratory study
Other: Permethrin higher dose — A fabric scarf, impregnated with the insecticide permethrin (m-Phenoxybenzyl)-cis,trans-3-(2,2-dichlorovinyl)-2,2-dimethylcyclopropanecarboxylate) that has contact irritancy/spatial repellency. Dose appropriate to children more than 20 kg.
  Arms: Field study: Permethrin higher dose; Laboratory study

SUMMARY:
Musca sorbens, a fly that feeds from ocular and nasal discharge on humans, is thought to be the vector of trachoma. We are developing methods of fly control that specifically target this species, in the hope of interrupting Ct transmission. To our knowledge, the use of commercially available insect repellents has never been tested for prevention of Musca sorbens fly-eye contact (i.e. nuisance and landing in the peri-ocular area). Given the likely necessity for prolonged and/or high frequency fly-eye contact for Ct transmission, the reduction of these contacts through the use of fly repellents presents an exciting opportunity for disease control. Here we propose a within-subject, non-masked, trial of the use of commercially available insect repellents against Musca sorbens, with two consecutive participant groups in the laboratory and in the field, and a primary endpoint of measuring the protective efficacy of each repellent product. Repellent products will be chosen from: DEET (N,N-diethyl-3-methylbenzamide), IR3535 (3-[N-butyl-N-acetyl]-aminopropionic acid ethyl ester), Picaridin (2-(2-hydroxyethyl)-1-piperidinecarboxylic acid 1-methylpropyl ester); PMD (para-Menthane-3,8-diol) or permethrin (m-Phenoxybenzyl)-cis,trans-3-(2,2-dichlorovinyl)-2,2-dimethylcyclopropanecarboxylate). Products tested will be either (1) topical repellents, or (2) in long-lasting, plastic formulations of repellents that can be worn on the body (wearable repellent technologies). The insect repellent synergist Vanillin (4-Hydroxy-3-methoxybenzaldehyde) may be added to the long-lasting plastic formulations, to improve the duration of protection.

DETAILED DESCRIPTION:
Introduction

Trachoma

Trachoma, a Neglected Tropical Disease (NTD), is the commonest infectious cause of blindness globally, affecting some of the world's poorest communities. Trachoma is caused by repeated ocular infection with the bacterium Chlamydia trachomatis (Ct). Active trachoma begins in childhood with recurrent episodes of follicular conjunctivitis (TF). Chronic inflammation results in immunologically mediated conjunctival scarring and in-turned eyelashes scratching the eye: trichiasis. Eventually sight is lost from irreversible corneal opacification.

Trachoma is currently endemic in 42 countries. The latest estimates from the Global Trachoma Mapping Programme (GTMP) suggest that 180 million people live in trachoma endemic areas and 3.2 million people have trachomatous trichiasis. Around 2.2 million people are visually impaired, of whom 1.2 million are blind. More than 80% of the burden of active trachoma is concentrated in 14 countries, mainly in the Sahel of West Africa and savannahs of East and Central Africa, where water supplies are often scarce.

Trachoma in Ethiopia

Ethiopia is working towards eliminating trachoma by 2020 and began implementing the SAFE strategy as part of national policy in 2003. This has focused on the provision of improved trichiasis surgery, mass drug administration (MDA) and the distribution of public health messages by radio, video, and printed material. From 2001-2015 more than one million trichiasis surgeries were performed, over 170 million doses of azithromycin were given through MDA and more than 24 million latrines were built. Despite these encouraging efforts, trachoma remains a public health problem in many regions of the country, and the burden of disease is far above the elimination targets set by the World Health Organisation (WHO). In many of these communities, despite seven years of annual or biannual high-coverage MDA, the prevalence of TF remains well above threshold for continuing MDA. Data on Ct prevalence after repeated rounds of MDA in hyperendemic settings such as Ethiopia, indicate that reliable long-term control is not consistently achieved, with gradual re-emergence of infection being typical.

Flies and Trachoma

Flies are likely to contribute to Ct transmission in some locations. The three members of the species complex Musca sorbens live in close association with humans across the Old World tropics and sub-tropics, Asia, the Pacific Islands and Australasian regions. The African species, M. sorbens and Musca biseta, are collectively known as The Bazaar fly, but all are also known as 'face flies', because of their habit of aggressively visiting the face to obtain the protein and liquid found in ocular and nasal secretions. When M. sorbens flies visit the face to feed, they can pick up Ct and transfer it on their bodies to another person. This is called mechanical transmission. Sometimes the house fly, Musca domestica, will also display eye-seeking behaviour, but across most trachoma-endemic regions, the vast majority of fly-eye contacts are made by M. sorbens. As well as transmitting trachoma, M. sorbens has been found to harbour enteric pathogens. In communities without adequate sanitation such as pit latrines, filth flies including M. sorbens have direct access to faecal breeding sites in the form of open defection. Here, they contact diarrhoea-causing pathogens, and subsequent contact to children's faces, or contamination of eating surfaces, can lead to pathogen transmission.

Ct can be cultured from guts and limbs of M. domestica fed on Ct-infected egg yolk. Using a tightly controlled guinea pig trachoma model, Chlamydia psittaci was transmitted by flies from infected to uninfected eyes. Infection was established consistently if the time between flies feeding on infected guinea pig ocular secretions and being exposed to uninfected guinea pigs was under one hour. Other, circumstantial, evidence suggests that flies contribute to the transmission of trachoma. In randomised controlled trials, significantly decreasing the M. sorbens population through long-term insecticide spraying led to decreases in the prevalence of clinical signs of active trachoma (infection not tested). However, azithromycin MDA combined with intensive insecticide spraying in other regions had no effect. Multiple transmission routes complicate trachoma epidemiology, and the extent to which flies contribute to transmission must also be dependent on local factors such as fly seasonality, abundance and local environmental factors that influence fly population dynamics. Two studies tested M. sorbens caught leaving faces of Ethiopian children for Ct by polymerase chain reaction (PCR); 15-23% of flies were positive. In The Gambia, Ct positive flies were also caught from children's faces. These data strongly suggest M. sorbens is a vector of trachoma, however, its relative importance probably varies by setting. Although it is probable that flies are involved in transmission, this pathway is poorly understood.

Olfactory cues have been exploited for monitoring and control of vector populations for many years, through the deployment of odour-baited traps. However, in recent years the use of such traps for population suppression of disease vectors has received increased attention, and recently the potential of these methods for malaria control was empirically demonstrated for the first time. One of the most long-standing and established examples of the use of odour-baited traps is the control of tsetse flies and Human African Trypanosomiasis in East Africa.

The investigators have recently conducted field studies in Oromia, Ethiopia, during Phase 1 and Phase 2 of the Stronger SAFE programme, designing a trap from locally sourced and cheaply available materials. The performance of this trap was tested, baited with a commercial lure, relative to several other commercially available fly traps and found to be superior. A major advantage of odour-baited trapping for fly control is that it is not associated with environmental impact concerns. This is in contrast to widespread insecticide spraying, which although has been shown to suppress fly populations very successfully, can be damaging to the environment.

Insect repellents are used world-wide to prevent nuisance biting by non-vector species, and to prevent disease transmission by vectors in disease-endemic regions. Although the use of plants with repellent qualities, either by burning leaves or presenting fresh foliage, is prevalent in many regions, commercially available topical repellents are rarely used by people in low-income and disease-endemic countries. This is because of cost, availability, and the impracticality of a product that requires repeat application. However, when use of insect repellents has been successfully adopted by communities, they have been found to be protective against malaria. Repellents have also been successfully used to control other arthropods of public health significance, including lice and the chigoe flea. A recent review of the evidence that topical insect repellents can be used to protect against clinical malaria or malaria infection found insufficient evidence, and called for better designed trials to generate higher-certainty evidence.

There is growing interest in the use of repellents as personal protection from disease transmission, particularly around the use of insecticide-treated clothing, which can repel biting insects. In these instances, the insecticide used has spatially repellent properties or is a contact irritant, which protects the individual user and the insecticides are not sprayed into the environment. Insecticide-treated clothing has been shown to provide protection from both malaria and leishmaniasis. Another study looked at the use of permethrin-treated headscarves for Afghan women in a Pakistani refugee camp, and found a reduction in the incidence of malaria in people under 20 years old. There is better evidence for the use of insecticide-treated clothing against malaria transmission, particularly advocated in areas where more evidence-based vector control strategies such as long-lasting insecticide-treated bed nets are not appropriate. Again, however, further high-quality studies are required to improve the efficacy evidence base.

Using the M. sorbens colony that the investigators have established at LSHTM, preliminary studies have been conducted that demonstrate M. sorbens are susceptible to most commercially available repellents. The investigators have found evidence that the insecticide permethrin has some spatial repellency to M. sorbens, if impregnated at safe doses into fabric scarves. In areas of high fly density, it is expected that the nuisance caused by these flies may allow such an intervention to be successful, as the immediate benefit of reduced face contact would encourage continued uptake of this intervention. Attractant (odour-baited trap) and repellent (commercially available repellents) technologies will be combined to create a "push-pull" strategy to reduce vector-host contact and attract flies to lethal odour-baited traps that will supress populations.

Research hypothesis

Commercially available insect repellent products can be used to decrease contact to the face, particularly the eyes, nose and mouth, by the eye-seeking fly Musca sorbens. The protection afforded by insect repellents will prevent transmission of Chlamydia trachomatis by infected flies, as well as reducing the nuisance caused by this species.

ELIGIBILITY:
Laboratory trial eligibility criteria

1. Participant is aged > 18 years and < 65 years and in good health
2. Participant has a good understanding of the procedures of the study and agrees to abide to these procedures
3. Participant is able to communicate well with the investigator, and attend the laboratory for all aspects of the laboratory studies
4. Participant has no known adverse reactions, or evidence at screening of adverse reactions, to the commercially available repellents DEET, PMD, IR3535, Picaridin or Permethrin, or to Vanilla
5. Participant has no known history of skin allergies or hypersensitivity to topical creams
6. Participant agrees to a pre-trial skin reactivity test for all the repellents that will be used in the trial
7. If in the event of the participant experiencing an adverse reaction to a repellent during the trial, the participant agrees to inform his/her general practitioner and seek appropriate treatment if necessary
8. Participant is willing to allow laboratory-reared Musca sorbens flies to land and crawl on their arm, during the modified arm-in-cage assay, for periods of up to ten minutes at a time
9. Participant agrees not to use any perfumed or scented product, including bathing products, for a 24-hour period before each laboratory session
10. Participant has signed informed consent
11. Participant is not a smoker, and will agree to refraining from smoking for the 12 hours before each laboratory trial

Field trial eligibility criteria

1. Participant lives in the designated study site
2. Participating households must be within a one-hour drive of Feya General Hospital
3. Participant considers themselves to be in good health, as does the parent or guardian
4. Participant is aged > 3 years and < 12 years
5. Participant has a good understanding of the procedures of the study and agrees to abide to these procedures
6. The parent or guardian of the participant has a good understanding of the procedures of the study and agrees to abide to these procedures
7. Participant is able to communicate well with the investigator or fieldworker who is conducting the study
8. Participant has no known adverse reactions to the commercially available repellents DEET, PMD, IR3535, Picaridin or Permethrin, or to Vanilla
9. Participant has no known history of skin allergies or hypersensitivity to topical creams
10. Participant agrees to a pre-trial skin reactivity test for all the repellents that will be used in the trial
11. If in the event of the participant experiencing an adverse reaction to a repellent during the trial, the participant can request medical advice from the Stronger-SAFE field team nurses if they wish
12. Participant is willing to sit still on a chair outside their house, for sequential periods of up to ten minutes, allowing wild fly contact and landing on the body and face, as much as possible without disturbing fly behaviour
13. Participant agrees not to use any perfumed or scented product, including bathing products, for a 24-hour period before each laboratory session
14. Able and willing to give fully informed assent
15. The parent or guardian has signed informed consent

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Protective Efficacy (PE) | 2 months
  The protection (protective efficacy, p) afforded by a repellent product will be presented as a percentage. p will be estimated by comparing fly-arm contact duration and fly-eye contact frequency, in laboratory and field trials respectively, after application (or wearing) of the repellent product to that during the control period.
Complete Protection Time (CPT) | 3 months
  Median CPT will be estimated in stage two ('persistence') laboratory trials only, for those repellents that demonstrated more than 30 % PE. The complete protection time for a specific dose will be estimated as the time elapsed until the first fly landing on the arm in each replicate, and based on repeat estimates of CPT, the mCPT will be estimated using a Kaplan-Meier function.

CONTACTS AND LOCATIONS:
Locations (2):
- Fred Hollows Foundation, Addis Ababa, Ethiopia
- London School of Hygiene and Tropical Medicine, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Formal reports will be written for the Ethiopian Federal and Regional health authority and the Federal Ministry of Science and Technology (FMOST). Reports will also be prepared for the Wellcome Trust and The Fred Hollows Foundation (Ethiopia and UK).
  To ensure operational uptake of the findings of the studies, we intend to present these data at the annual National Trachoma Task Force and NTD Research Symposium (Ethiopia). Additionally, we will present this research at the annual Trachoma Scientific Informal Workshop prior to the WHO GET2020 Alliance meeting. Scientific results will be published in Open Access in peer-reviewed journals and presented at relevant international conferences.
  The Sensitisation/Community Liaison Team will disseminate the results of the study to the study community in community dialogues and radio broadcasts in conjunction with The Fred Hollows Foundation Ethiopia Communications Team.

REFERENCES:
- [Background] Banks SD, Murray N, Wilder-Smith A, Logan JG. Insecticide-treated clothes for the control of vector-borne diseases: a review on effectiveness and safety. Med Vet Entomol. 2014 Aug;28 Suppl 1:14-25. doi: 10.1111/mve.12068. Epub 2014 Jun 10. PMID 24912919
- [Background] Bell, M.J. (2018) The impact of latrine construction on densities and pathogen infection rates of synanthropic flies and Culex quinquefasciatus mosquitoes in Odisha, India. PhD thesis.
- [Background] Burgess, I. (1993) The function of a repellent in head louse control. The Pharmaceutical Journal. 15, 674-675.
- [Background] Emerson PM, Bailey RL, Mahdi OS, Walraven GE, Lindsay SW. Transmission ecology of the fly Musca sorbens, a putative vector of trachoma. Trans R Soc Trop Med Hyg. 2000 Jan-Feb;94(1):28-32. doi: 10.1016/s0035-9203(00)90427-9. PMID 10748893
- [Background] Emerson PM, Bailey RL, Walraven GE, Lindsay SW. Human and other faeces as breeding media of the trachoma vector Musca sorbens. Med Vet Entomol. 2001 Sep;15(3):314-20. doi: 10.1046/j.0269-283x.2001.00318.x. PMID 11583450
- [Background] Emerson PM, Lindsay SW, Alexander N, Bah M, Dibba SM, Faal HB, Lowe KO, McAdam KP, Ratcliffe AA, Walraven GE, Bailey RL. Role of flies and provision of latrines in trachoma control: cluster-randomised controlled trial. Lancet. 2004 Apr 3;363(9415):1093-8. doi: 10.1016/S0140-6736(04)15891-1. PMID 15064026
- [Background] European Commission (2014) Assessment Report: Permethrin. Available at: http://dissemination.echa.europa.eu/Biocides/ActiveSubstances/1342-18/1342-18_Assessment_Report.pdf
- [Background] Faulde M, Uedelhoven W. A new clothing impregnation method for personal protection against ticks and biting insects. Int J Med Microbiol. 2006 May;296 Suppl 40:225-9. doi: 10.1016/j.ijmm.2006.01.008. Epub 2006 Mar 9. PMID 16524779
- [Background] Feldmeier H, Kehr JD, Heukelbach J. A plant-based repellent protects against Tunga penetrans infestation and sand flea disease. Acta Trop. 2006 Oct;99(2-3):126-36. doi: 10.1016/j.actatropica.2006.05.013. Epub 2006 Sep 29. PMID 17010927
- [Background] Forsey T, Darougar S. Transmission of chlamydiae by the housefly. Br J Ophthalmol. 1981 Feb;65(2):147-50. doi: 10.1136/bjo.65.2.147. PMID 7459318
- [Background] Heng S, Durnez L, Gryseels C, Van Roey K, Mean V, Uk S, Siv S, Grietens KP, Sochantha T, Coosemans M, Sluydts V. Assuring access to topical mosquito repellents within an intensive distribution scheme: a case study in a remote province of Cambodia. Malar J. 2015 Nov 24;14:468. doi: 10.1186/s12936-015-0960-4. PMID 26597653
- [Background] Hill N, Lenglet A, Arnez AM, Carneiro I. Plant based insect repellent and insecticide treated bed nets to protect against malaria in areas of early evening biting vectors: double blind randomised placebo controlled clinical trial in the Bolivian Amazon. BMJ. 2007 Nov 17;335(7628):1023. doi: 10.1136/bmj.39356.574641.55. Epub 2007 Oct 16. PMID 17940319
- [Background] Homan T, Hiscox A, Mweresa CK, Masiga D, Mukabana WR, Oria P, Maire N, Pasquale AD, Silkey M, Alaii J, Bousema T, Leeuwis C, Smith TA, Takken W. The effect of mass mosquito trapping on malaria transmission and disease burden (SolarMal): a stepped-wedge cluster-randomised trial. Lancet. 2016 Sep 17;388(10050):1193-201. doi: 10.1016/S0140-6736(16)30445-7. Epub 2016 Aug 9. PMID 27520594
- [Background] Lee S, Alemayehu W, Melese M, Lakew T, Lee D, Yi E, Cevallos V, Donnellan C, Zhou Z, Chidambaram JD, Gaynor BD, Whitcher JP, Lietman TM. Chlamydia on children and flies after mass antibiotic treatment for trachoma. Am J Trop Med Hyg. 2007 Jan;76(1):129-31. PMID 17255240
- [Background] Maia MF, Kliner M, Richardson M, Lengeler C, Moore SJ. Mosquito repellents for malaria prevention. Cochrane Database Syst Rev. 2018 Feb 6;2(2):CD011595. doi: 10.1002/14651858.CD011595.pub2. PMID 29405263
- [Background] Massue DJ, Moore SJ, Mageni ZD, Moore JD, Bradley J, Pigeon O, Maziba EJ, Mandike R, Kramer K, Kisinza WN, Overgaard HJ, Lorenz LM. Durability of Olyset campaign nets distributed between 2009 and 2011 in eight districts of Tanzania. Malar J. 2016 Mar 18;15:176. doi: 10.1186/s12936-016-1225-6. PMID 26993981
- [Background] Miller K, Pakpour N, Yi E, Melese M, Alemayehu W, Bird M, Schmidt G, Cevallos V, Olinger L, Chidambaram J, Gaynor B, Whitcher J, Lietman T. Pesky trachoma suspect finally caught. Br J Ophthalmol. 2004 Jun;88(6):750-1. doi: 10.1136/bjo.2003.038661. PMID 15148205
- [Background] Moore SJ, Hill N, Ruiz C, Cameron MM. Field evaluation of traditionally used plant-based insect repellents and fumigants against the malaria vector Anopheles darlingi in Riberalta, Bolivian Amazon. J Med Entomol. 2007 Jul;44(4):624-30. doi: 10.1603/0022-2585(2007)44[624:feotup]2.0.co;2. PMID 17695017
- [Background] Orsborne J, DeRaedt Banks S, Hendy A, Gezan SA, Kaur H, Wilder-Smith A, Lindsay SW, Logan JG. Personal Protection of Permethrin-Treated Clothing against Aedes aegypti, the Vector of Dengue and Zika Virus, in the Laboratory. PLoS One. 2016 May 17;11(5):e0152805. doi: 10.1371/journal.pone.0152805. eCollection 2016. PMID 27187593
- [Background] Paru R, Hii J, Lewis D, Alpers MP. Relative repellency of woodsmoke and topical applications of plant products against mosquitoes. P N G Med J. 1995 Sep;38(3):215-21. PMID 9522861
- [Background] Richards SL, Balanay JAG, Harris JW, Banks VM, Meshnick S. Residual Effectiveness of Permethrin-Treated Clothing for Prevention of Mosquito Bites Under Simulated Conditions. J Environ Health. 2017 Apr;79(8):8-15. PMID 29148650
- [Background] Rowland M, Durrani N, Hewitt S, Mohammed N, Bouma M, Carneiro I, Rozendaal J, Schapira A. Permethrin-treated chaddars and top-sheets: appropriate technology for protection against malaria in Afghanistan and other complex emergencies. Trans R Soc Trop Med Hyg. 1999 Sep-Oct;93(5):465-72. doi: 10.1016/s0035-9203(99)90341-3. PMID 10696399
- [Background] Schwalfenberg S, Witt LH, Kehr JD, Feldmeier H, Heukelbach J. Prevention of tungiasis using a biological repellent: a small case series. Ann Trop Med Parasitol. 2004 Jan;98(1):89-94. doi: 10.1179/000349804225003091. No abstract available. PMID 15000736
- [Background] Sholdt LL, Schreck CE, Mwangelwa MI, Nondo J, Siachinji VJ. Evaluations of permethrin-impregnated clothing and three topical repellent formulations of deet against tsetse flies in Zambia. Med Vet Entomol. 1989 Apr;3(2):153-8. doi: 10.1111/j.1365-2915.1989.tb00493.x. PMID 2519659
- [Background] Sluydts V, Durnez L, Heng S, Gryseels C, Canier L, Kim S, Van Roey K, Kerkhof K, Khim N, Mao S, Uk S, Sovannaroth S, Grietens KP, Sochantha T, Menard D, Coosemans M. Efficacy of topical mosquito repellent (picaridin) plus long-lasting insecticidal nets versus long-lasting insecticidal nets alone for control of malaria: a cluster randomised controlled trial. Lancet Infect Dis. 2016 Oct;16(10):1169-1177. doi: 10.1016/S1473-3099(16)30148-7. Epub 2016 Jun 29. PMID 27371977
- [Background] Soto J, Medina F, Dember N, Berman J. Efficacy of permethrin-impregnated uniforms in the prevention of malaria and leishmaniasis in Colombian soldiers. Clin Infect Dis. 1995 Sep;21(3):599-602. doi: 10.1093/clinids/21.3.599. PMID 8527550
- [Background] West SK, Emerson PM, Mkocha H, McHiwa W, Munoz B, Bailey R, Mabey D. Intensive insecticide spraying for fly control after mass antibiotic treatment for trachoma in a hyperendemic setting: a randomised trial. Lancet. 2006 Aug 12;368(9535):596-600. doi: 10.1016/S0140-6736(06)69203-9. PMID 16905024
- [Background] World Health Organization (2017) How to design vector control efficacy trials: Guidance on phase III vector control field trial design provided by the Vector Control Advisory Group.
- [Derived] Robinson A, Gomes LRO, Abdurahman OS, Alemayehu W, Shuka G, Melese E, Guye M, Legesse D, Elias E, Temam K, Koro KH, Adugna D, Seife F, Aga MA, Sarah V, Lambert SM, Walker SL, Habtamu E, Solomon AW, Last A, Macleod D, Burton MJ, Logan JG. Evaluation of the efficacy of insecticide-treated scarves to protect children from the trachoma vector Musca sorbens (Diptera: Muscidae): A phase II randomised controlled trial in Oromia, Ethiopia. EClinicalMedicine. 2022 Jun 8;49:101487. doi: 10.1016/j.eclinm.2022.101487. eCollection 2022 Jul. PMID 35747196

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT03813069/Prot_SAP_000.pdf